CLINICAL TRIAL: NCT01863095
Title: Use of Exercise to Reduce Young Adult Marijuana Use: There is an App for That
Brief Title: An Exercise App to Reduce Young Adults' MJ Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, R. Lorraine Collins, Ph.D., Professor, Community Health and Health Behavior, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34DA035358 (NIH)
Record Dates: First submitted 2013-05-21; First posted 2013-05-27 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Marijuana Smoking
MeSH Terms: conditions — Marijuana Smoking | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): MJ users assigned to this condition will participate in 4 individualized intervention sessions that are based on Motivational Interviewing principles. They will receive personalized feedback on their MJ use and will be provided a smart phone app on which they report their MJ use episodes, which also is designed to promote the use of exercise/physical activity as an alternative to MJ use. Level of Physical activity will be measured using accelerometers.
  Interventions: Behavioral: Personalized Feedback and Exercise
- Personalized Feedback only (Active Comparator): MJ users assigned to this condition will participate in 4 individualized intervention sessions that are based on Motivational Interviewing principles. They will only receive personalized feedback on their MJ use.
  Interventions: Behavioral: Personalized Feedback and Exercise

INTERVENTIONS:
Behavioral: Personalized Feedback and Exercise

SUMMARY:
Currently, marijuana (MJ) is the most popular illicit drug, but there are few effective interventions to help young adults (age 18 to 25 years) to reduce their MJ intake. In this study, we will develop and initially test a smart phone app designed to promote exercise/physical activity as a positive alternative to MJ use. The app will be tested in an efficacy study in which MJ users are randomly to either receive personalized feedback about MJ use + use the exercise app or personalized feedback only. The results will contribute to knowledge about exercise/physical activity as a strategy for reducing young adults' MJ use and problems.

DETAILED DESCRIPTION:
Currently, marijuana (MJ) is the most popular illicit drug, with prevalence studies indicating increasing use among young adults (Johnston et al., 2011). Even so, there are few effective interventions to help MJ users reduce their intake to avoid negative consequences, including MJ dependence. The investigators propose a Stage 1 efficacy study to develop and initially test an innovative intervention to reduce MJ use among young adults who regularly use MJ (> 3 episodes/week). The intervention includes elements from the Marijuana Check-Up (MCU; Stephens et al., 2007), a MI-based brief intervention that has shown promise for reducing MJ use. It also incorporates findings from our ongoing research, which suggest that exercise/physical activity (PA) has potential as a positive alternative to MJ use. The investigators research also has shown that short (i.e., 10 minute) bouts of moderate or intense exercise reduce craving/urges to use MJ. Exercise interventions have successfully reduced use of licit substances, such as tobacco (e.g., Marcus et al., 2005) and alcohol (e.g., Brown et al., 2009), but have not been adequately tested for MJ use. The two aims of this R34 application are: 1) To develop an intervention that consists of four, 60-minute, in-person sessions composed of MCU content (e.g., personalized feedback, MI) as well as a smart phone application (app) that promotes exercise/physical activity (EA) as an alternative to MJ use. The EA, which will be designed to specifically appeal to young adults, will provide a readily-accessible, flexible, and convenient platform for personalized information and reminders that promote exercise/PA as a positive alternative to MJ use in ongoing daily life. 2) To conduct a pilot/efficacy study of the 4-week MCU+EA intervention vs. a MCU-only control condition. The investigators will use urn randomization to assign emerging/young-adult MJ users (N = 40) to the two conditions. During the 1-week baseline, 4-week intervention phase, and 1-, 3-, and 6-month follow-ups, all participants will use the smart phone app to provide real-time data on MJ-related variables and wear accelerometers to provide PA data. Multilevel modeling will be used to test our hypothesis that the MCU+EA intervention, compared to MCU-only control, will produce greater decreases in quantity and frequency of MJ use (and related MJ problems) at post-intervention and at each follow-up. Multilevel modeling also will be used to explore the real-time data to examine the role of variables such as urge/craving for MJ, social factors, and dosage of PA in the reduction of the quantity and frequency of MJ use. This Stage 1 study is unique and innovative in its development and use of a smart phone app to promote and evaluate exercise/PA as a positive alternative to MJ use in daily life. It includes cutting-edge technology (e.g., accelerometers, smart phone app) for real-time assessments. This research will make significant contributions to the limited knowledge of exercise/PA as a strategy for reducing MJ use and related problems among emerging and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Regular Marijuana user interested in cutting down on marijuana use
* Body Mass Index < 30

Exclusion Criteria:

* Pregnant or planning to become pregnant
* No legal problems
* No substance abuse diagnosis
* No history of substance abuse treatment
* Medical contraindications to engaging in exercise
* Psychological distress or psychiatric treatment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Physical Activity | Change in exercise at 1 month, 3 months, and 6 months after interventionts
  Counts based on data collected by accelerometers.
Substance Use | Change in marijuana use at 1 month, 3 months, and 6 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: R Lorraine Collins, Ph.D., Principal Investigator — State University of New York at Buffalo
Locations (1):
- Center for Health Research, Buffalo, New York, United States